CLINICAL TRIAL: NCT07320222
Title: A Coordinated Approach to Peri-operative Rehabilitation to Enhance Outcomes in Melanoma: the CARE-Melanoma Pilot Randomized Controlled Trial
Brief Title: CARE-Melanoma Trial
Acronym: CARE-Melanoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CARE-Melanoma
Record Dates: First submitted 2025-11-24; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Melanoma (Skin Cancer)
Keywords: rehabilitation; melanoma; peri-operative; pilot trial
MeSH Terms: conditions — Melanoma | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: This is a two group pilot randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARE Intervention Group (Experimental): This intervention group will include four peri-operative intervention sessions, the total intervention time will be approximately 4 months, with two of the intervention sessions will occur prior to surgery, and two occurring post-surgery. At the pre-surgery sessions individuals with receive education on the benefits of exercise pre-treatment, how to exercise safely, and be set up with a tailored exercise routine by a trained physiotherapist. They will set goals and action plans to work until their next session. At the post-surgery sessions patients will review their function with the same physiotherapist and again be provided tailored recommendations to maximize their function.
  Interventions: Other: Rehabilitation
- Usual Care (No Intervention): This group will receive usual care (no rehabilitation intervention).

INTERVENTIONS:
Other: Rehabilitation — Includes education on the benefit of exercise and how to exercise safely, rehabilitation to maximize strength, range of motion, and function, set up with a tailored exercise program by a trained physiotherapist or kinesiologist, goal setting and action planning.
  Arms: CARE Intervention Group

SUMMARY:
Melanoma, a serious skin cancer, is increasingly prevalent in Canada. Surgical intervention is essential but poses significant physical and emotional challenges. Rehabilitation is crucial for recovery, helping patients regain strength and confidence while addressing psychological needs. In Ontario, new neoadjuvant chemotherapy regimens are being introduced to improve outcomes by shrinking tumors before surgery. Despite advancements, pre-habilitation and early post-operative rehabilitation services for melanoma patients are currently lacking. This pilot trial aims to evaluate the feasibility and effectiveness of pre- and post-surgery rehabilitation strategies for melanoma patients. The purpose of this pilot trial is to determine the feasibility and preliminary effectiveness of a rehabilitation strategy for individuals with melanoma pre- and post-surgery.

DETAILED DESCRIPTION:
Melanoma, a serious skin cancer, is increasingly prevalent in Canada. Surgical intervention is essential but poses significant physical and emotional challenges. Rehabilitation is crucial for recovery, helping patients regain strength and confidence while addressing psychological needs. In Ontario, new neoadjuvant chemotherapy regimens are being introduced to improve outcomes by shrinking tumors before surgery. Despite advancements, pre-habilitation and early post-operative rehabilitation services for melanoma patients are currently lacking. This pilot trial aims to evaluate the feasibility and effectiveness of pre- and post-surgery rehabilitation strategies for melanoma patients. Participants in this study include individuals with a melanoma diagnosis who are scheduled to receive surgery after a neoadjuvant chemotherapy regime. Eligible potential participants will be referred to the study by their surgical oncologist or oncology care. Participants will be screened for eligibility by a research coordinator. Based on sample size calculations for pilot data, the investigators expect to recruit 30 participants for the study (15 in each group). Participants will be divided into two groups. The first group will include four peri-operative intervention sessions, the total intervention time will be approximately 4 months, with two of the intervention sessions occurring prior to surgery, and two occurring post-surgery. At the pre-surgery sessions participants with receive education on the benefits of exercise pre-treatment, how to exercise safely, and be set up with a tailored exercise routine by a trained physiotherapist. Participants will set goals and action plans to work until their next session. At the post-surgery sessions patients will review their function with the same physiotherapist and again be provided tailored recommendations to maximize their function. The second group will receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* melanoma diagnosis
* English speaking,
* adults (>18 years of age)
* scheduled to receive surgery after a neoadjuvant chemotherapy regime

Exclusion Criteria:

* <18 years of age
* are not undergoing neo-adjuvant chemotherapy
* self-report any chronic condition, cognitive impairment, or injury that would prevent them from participating independently in moderate intensity exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Retention rate | 4 months
  Retention rate is the number of individuals enrolled in the study who complete the intervention.

SECONDARY OUTCOMES:
Adherence rate | 4 months
  Adherence in this project will be assessed by adherence to the rehabilitation session (measured as %).
Recruitment rate | 4 months
  Recruitment rate is the percentage of eligible individuals approached for the study who enrol in the study.
Change in overall impairment score | 4 months
  Measured via the Edmonton Symptom Assessment Scale at baseline and 4 month follow-up. Minimum score: 0, Maximum score: 100 - higher scores represent higher levels of overall impairment.
Change in Physical Activity Level | 4 months
  Measured via the Godin Leisure Time Exercise Questionnaire at baseline and 4 month follow-up. Minimum score: 0, Maximum score: no max - higher scores represent higher levels of physical activity.
Change in functional mobility | 4 months
  Measured via the 30 second sit to stand at baseline and 4 month follow-up. Minimum score: 0, Maximum score: no max - higher scores represent higher levels of functional mobility.
Change in functional mobility | 4 months
  Measured via the six minute walk test at baseline and 4 month follow-up. Minimum score: 0, Maximum score: no max - higher scores represent higher levels of functional mobility.
Change in Grip Strength | 4 months
  Measured via the handheld dynamometer at baseline and 4 month follow-up
Change in quality of life | 4 months
  Measured via the Functional Assessment of Cancer Therapy (FACT)-Melanoma at baseline and 4 month follow-up. Minimum score: 0, Maximum score: 204 - higher scores represent higher levels of quality of life.
Change in perception of health status | 4 months
  Measured via the EQ-5D-3L VAS (no extended title) at baseline and 4 month follow-up. Minimum score: 0, Maximum score: 100 - higher scores represent higher perceptions of health status.
Medication use | 4 months
  Measured via a self-report scale at 4 month follow-up. Minimum score: 0 (no medication used), Maximum score: no maximum - higher scores represent higher use of medications.
Change in range of motion | 4 months
  Measured via the goniometer at baseline and 4 month follow-up

IPD SHARING:
Plan to Share IPD: No